CLINICAL TRIAL: NCT06643897
Title: Identification of Barriers and Facilitators of Implementation of the Out-of-Hospital Administration of the Long- Acting Combination Cabotegravir+Rilpivirina as an Optional Therapy in People Living With HIV From Spain.
Brief Title: Identification of Barriers and Facilitators of Implementation of the Out-of-Hospital Administration of the Long- Acting Combination Cabotegravir+Rilpivirina.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Substudy LA CAB+RPV
Record Dates: First submitted 2024-10-08; First posted 2024-10-16 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: HIV-1-infection
Keywords: barriers and facilitators; interview; long acting; out-of-hospital by implementation; cabotegravir + rilpivirine (CAB+RPV); HIV-1

STUDY DESIGN:
Intervention Model Description: The substudy is a transversal, one arm, multicentric study including the staff participating in the HOLA study, to identify the barriers and facilitators of implementation of the out-of-hospital administration of CAB+RPV LA following a qualitative descriptive design.
  All study staff who participate in the substudy will be interviewed through a 40-50 minute-qualitative interview
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Qualitative Interview (Other): All study staff who participate in the substudy will be interviewed through a 40-50 minute-qualitative interview.
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Other: Qualitative Interview — 40-50 minute-qualitative interview.

SUMMARY:
The study will identify the barriers and facilitators of implementation of the out-of-hospital administration of CAB+RPV LA from the point of view of staff participating in the study.

DETAILED DESCRIPTION:
This substudy will use a qualitative descriptive approach based on Consolidated Framework for Implementation Research (CFIR). Data will be collected using semi-structured interviews among HOLA staff participants until achieving data saturation. Data will be analyzed using Braun & Clarke's thematic analysis method.

ELIGIBILITY:
Inclusion Criteria:

1. Participation throughout the HOLA study until the moment of conducting the interviews and direct involvement in the study procedures in a significant way.
2. Homogeneous sample between the different roles participating in the study.
3. Participants who agree to participate in the substudy and sign the informed consent.

Exclusion Criteria: NONE

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Identify the barriers and facilitators of implementation of the out-of-hospital administration of CAB+RPV LA from the point of view of staff participating in the study. | after the first 6 months of participation in the study
  1. To assess barriers and facilitators of implementation of the out-of-hospital administration of CAB+RPV LA from the point of view of staff participating in the HOLA study, at any time after the first 6 months of participation in the study. These will be assessed through a 40-50 minute-qualitative interview created for the study, which references the following domains: adaptability to the intervention, consideration of the needs of patients, changes in infrastructure, implementation climate (need of change, compatibility), preparation for implementation (leadership engagement and resource availability), individual characteristics, need for external agents, main stakeholders, execution and final considerations.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Germans Trias I Pujol Hospital, Badalona, Barcelona
  - CAP Dr Robert, Barcelona
  - Centre de Salut Internacional i Malalties Transmissibles Drassanes - Vall d'Hebron, Barcelona
  - BCN CheckPoint, Barcelona
  - Hospital Vall D' Hebrón, Barcelona
  - Cs Leganitos, Málaga
  - Hospital Costa Del Sol, Málaga
  - Cs San Luis de Sabinillas, Málaga
  - Cs San Pedro de Alcántara, Málaga

REFERENCES:
- [Derived] Hernandez-Sanchez D, Leyva-Moral JM, Olalla J, Negredo E, On Behalf Of The Hola Study Group. Barriers and Facilitators of Implementation of the Non-Hospital-Based Administration of Long-Acting Cabotegravir Plus Rilpivirine in People with HIV: Qualitative Data from the HOLA Study. Viruses. 2025 Jul 16;17(7):993. doi: 10.3390/v17070993. PMID 40733609